CLINICAL TRIAL: NCT00721136
Title: Randomized Study of the Use of Warfarin During Pacemaker or ICD Implantation in Patients Requiring Long Term Anticoagulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NA_00011273
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-07

CONDITIONS: Bradycardia; Tachycardia; Atrial Fibrillation; Valvular Heart Disease
Keywords: bleeding; anticoagulation; pacemaker; implantable cardioverter-defibrillator; patients undergoing implantation of a pacemaker or defibrillator (ICD)"
MeSH Terms: conditions — Bradycardia; Tachycardia; Atrial Fibrillation; Heart Valve Diseases; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Moderate risk patients (afib, mechanical aortic valve) randomized to continue coumadin at their usual dose through the procedure.
  Interventions: Drug: continue warfarin through the procedure
- 2 (Active Comparator): Moderate risk patients randomized to hold their coumadin for 4-5 days prior to the procedure (to allow the INR to normalize).
  Interventions: Drug: Hold warfarin
- 3 (Experimental): High risk patients (mechanical mitral valve, prior stroke, current deep vein thrombosis, hypercoagulable syndrome) randomized to continue coumadin at the usual dose through the procedure.
  Interventions: Drug: continue warfarin through the procedure
- 4 (Active Comparator): High risk patients randomized to holding coumadin for 4-5 days and using "bridging" anticoagulation with heparin while the coumadin is held.
  Interventions: Drug: Warfarin held with heparin transition.

INTERVENTIONS:
Drug: continue warfarin through the procedure — The usual dose of warfarin (resulting in a therapeutic INR) is taken throughout the peri-procedural period.
  Arms: 1; 3
Drug: Hold warfarin — For moderate risk patients, warfarin will be held for 4-5 days prior to the procedure.
  Arms: 2
Drug: Warfarin held with heparin transition. — For high risk patients, warfarin is held for 4-5 days prior to the procedure and heparin is given to provide anticoagulation while the INR is subtherapeutic.
  Arms: 4

SUMMARY:
Patients requiring long term anticoagulation often undergo transition of their warfarin to heparin in anticipation of invasive surgical procedures such as pacemaker or ICD implantation. This may require inpatient hospitalization several days prior to and after the procedure, potentially increasing medical costs and patient inconvenience. Patients undergoing such a process are initiated on heparin while their INRs drift to normal levels. Immediately prior to surgery, heparin is discontinued and restarted several hours after the procedure. Unfortunately, this process has resulted in a high incidence of surgical wound hematomas and other bleeding complications often requiring longer periods of discontinued anticoagulation or repeat surgical exploration. Previous investigators have tried to reduce the incidence of wound hematomas by prolonging the time from surgical wound closure to the reinitiation of heparin. A small randomized trial demonstrated that there was no significant difference in the incidence of wound hematomas whether heparin was started 6 hours or 24 hours after surgery (J Am Coll Cardiology 2000;35:1915-8). This has led many investigators to perform pacemaker and ICD implantation without reversal of warfarin therapy. A recent retrospective observational study demonstrated that the incidence of wound hematomas in patients with an INR of 2.6 was no different than patients with an INR of 1.5 (PACE 2004;27:358-60). Furthermore, a more recent, larger retrospective observational study reported in abstract form at the recent Heart Rhythm Society Annual 2007 Scientific Meeting demonstrated that not only is performing pacemaker and ICD implantations safe without reversing warfarin anticoagulation, but the incidence of wound hematomas is significantly smaller as compared to the strategy of reversing warfarin and initiating periprocedural heparin.

Given these findings, the hypothesis of this randomized study is that pacemaker and ICD implantation while fully anticoagulated on warfarin therapy is safe. Findings from this study will have significant implications on the clinical practice of pacemaker or ICD implantation in this patient population given that no randomized study on this subject has been performed to date.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for clinically indicated permanent pacemaker or implantable cardioverter-defibrillator
* currently on chronic warfarin therapy

Exclusion Criteria:

* unwilling to participate in trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Cheng, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Howard County General Hospital, Columbia, Maryland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients from each treatment arm were excluded from the analysis. Three of these patients withdrew after being told of the treatment assignment, and one patient's procedure was cancelled owing to need for a left ventricular assist device.
Groups:
- Moderate Risk Continuing Warfarin (Coumadin): Moderate risk patients (afib, mechanical aortic valve) randomized to continue coumadin at their usual dose through the procedure.
  These patients continue warfarin through the procedure : The usual dose of warfarin (resulting in a therapeutic INR) is taken throughout the peri-procedural period.
- Moderate Risk Holding Warfarin (Coumadin): Moderate risk patients randomized to hold their coumadin for 4-5 days prior to the procedure (to allow the INR to normalize).
  These patients hold warfarin : For moderate risk patients, warfarin will be held for 4-5 days prior to the procedure.
- High Risk Continuing Warfarin (Coumadin): High risk patients (mechanical mitral valve, prior stroke, current deep vein thrombosis, hypercoagulable syndrome) randomized to continue warfarin at the usual dose through the procedure.
  These patients continue warfarin through the procedure : The usual dose of warfarin (resulting in a therapeutic INR) is taken throughout the peri-procedural period.
- High Risk Holding Warfarin (Coumadin): These high risk patients randomized to holding warfarin for 4-5 days and using a heparin transition for bridging.
Period: Overall Study
Arm/Group | Moderate Risk Continuing Warfarin (Coumadin) | Moderate Risk Holding Warfarin (Coumadin) | High Risk Continuing Warfarin (Coumadin) | High Risk Holding Warfarin (Coumadin)
Started | 42 | 42 | 8 | 8
Completed | 42 | 42 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moderate Risk Continuing Warfarin: Moderate risk patients (afib, mechanical aortic valve) randomized to continue coumadin at their usual dose through the procedure.
  These patients continue warfarin through the procedure : The usual dose of warfarin (resulting in a therapeutic INR) is taken throughout the peri-procedural period.
- Moderate Risk Holding Warfarin: Moderate risk patients randomized to hold their coumadin for 4-5 days prior to the procedure (to allow the INR to normalize).
  These patients hold warfarin : For moderate risk patients, warfarin will be held for 4-5 days prior to the procedure.
- High Risk Continuing Warfarin: High risk patients (mechanical mitral valve, prior stroke, current deep vein thrombosis, hypercoagulable syndrome) randomized to continue coumadin at the usual dose through the procedure.
  These patients continue warfarin through the procedure : The usual dose of warfarin (resulting in a therapeutic INR) is taken throughout the peri-procedural period.
- High Risk Holding Warfarin: These high risk patients randomized to holding coumadin for 4-5 days and using a heparin transition for bridging.
- Total: Total of all reporting groups
Arm/Group | Moderate Risk Continuing Warfarin | Moderate Risk Holding Warfarin | High Risk Continuing Warfarin | High Risk Holding Warfarin | Total
Number analyzed (Participants) | 42 | 42 | 8 | 8 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 4 | 4 | 50
  >=65 years | 21 | 21 | 4 | 4 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (11.4) | 68.8 (11.7) | 72.9 (11.4) | 68.8 (11.7) | 71.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 2 | 2 | 42
  Male | 24 | 22 | 6 | 6 | 58
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 8 | 8 | 100

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Complication
Description: Significant bleeding was defined as extracardiac bleeding or pocket hematomas that required additional intervention and/or temporary discontinuation of anticoagulation therapy.
Time Frame: 30 days
Population: Baseline characteristics of both groups were well matched except that patients randomized to warfarin discontinuation were more obese (P = .024).
Measure: Number; unit: participants
Groups:
- Moderate Risk Continuing Warfarin: Moderate risk patients (afib, mechanical aortic valve) randomized to continue coumadin at their usual dose through the procedure.
  These patients continue warfarin through the procedure:The usual dose of warfarin (resulting in a therapeutic INR) is taken throughout the peri-procedural period.
- High Risk Continuing Warfarin: High risk patients (mechanical mitral valve, prior stroke, current deep vein thrombosis, hypercoagulable syndrome) randomized to continue warfarin at the usual dose through the procedure.
  These patients continue warfarin through the procedure: The usual dose of warfarin (resulting in a therapeutic INR) is taken throughout the peri-procedural period.
- High Risk Holding Warfarin: These high risk patients randomized to holding warfarin for 4-
Arm/Group | Moderate Risk Continuing Warfarin | Moderate Risk Holding Warfarin | High Risk Continuing Warfarin | High Risk Holding Warfarin
Number analyzed (Participants) | 39 | 41 | 7 | 8
participants | 0 | 2 | 0 | 2
Statistical Analysis 1: Comparison: Moderate Risk Continuing Warfarin vs Moderate Risk Holding Warfarin; Continuous variables were expressed as mean ± standard deviation and analyzed using Student's t-test and Mann-Whitney U-test in cases of nonparametric distribution. Categorical variables were expressed as numbers or percentages and analyzed with two-tailed Fisher's exact test or χ2-test as appropriate. Data were analyzed on an intention-to-treat basis using STATA 10.1 (College Station, TX). A two-tailed alpha of 0.05 was considered statistically significant; Test type: Other; Continuous variables were expressed as mean ± standard deviation and analyzed using Student's t-test and Mann-Whitney U-test in cases of nonparametric distribution. Categorical variables were expressed as numbers or percentages and analyzed with two-tailed Fisher's exact test or χ2-test as appropriate. Data were analyzed on an intention-to-treat basis using STATA 10.1 (College Station, TX). A two-tailed alpha of 0.05 was considered statistically significant

2. Primary Outcome: Thromboembolic Events
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Moderate Risk Continuing Warfarin (Coumadin) | Moderate Risk Holding Warfarin (Coumadin) | High Risk Continuing Warfarin (Coumadin) | High Risk Holding Warfarin (Coumadin)
Number analyzed (Participants) | 39 | 41 | 7 | 8
participants | 0 | 1 | 0 | 0

3. Primary Outcome: Anticoagulant Related Complications
Description: Defined as warfarin induced skin necrosis or heparin-induced thrombocytopenia
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Moderate Risk Continuing Warfarin (Coumadin) | Moderate Risk Holding Warfarin (Coumadin) | High Risk Continuing Warfarin (Coumadin) | High Risk Holding Warfarin (Coumadin)
Number analyzed (Participants) | 39 | 41 | 7 | 8
participants | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Groups:
- High Risk Continuing Warfarin: High risk patients (mechanical mitral valve, prior stroke, current deep vein thrombosis, hypercoagulable syndrome) randomized to continue warfarin at the usual dose through the procedure.
- High Risk Holding Warfarin: These patients continue warfarin through the procedure : The usual dose of warfarin (resulting in a therapeutic INR) is taken throughout the peri-procedural period.
  These high risk patients randomized to holding warfarin for 4-5 days and using a heparin transition for bridging.
Arm/Group | Moderate Risk Continuing Warfarin | Moderate Risk Holding Warfarin | High Risk Continuing Warfarin | High Risk Holding Warfarin
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/42 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/42 | 1/42 | 0/8 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Risk Continuing Warfarin (N=42) | Moderate Risk Holding Warfarin (N=42) | High Risk Continuing Warfarin (N=8) | High Risk Holding Warfarin (N=8)
Transient Ischemic Attack (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Risk Continuing Warfarin (N=42) | Moderate Risk Holding Warfarin (N=42) | High Risk Continuing Warfarin (N=8) | High Risk Holding Warfarin (N=8)
Pocket Hematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pericardial Effusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Evaluation period was limited to 4-6 weeks after implantation and mean INR levels in the warfarin continuation group did not reach levels above 2.5. This was a single center trial with experienced electrophysiologists using a common technique.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No